CLINICAL TRIAL: NCT01912482
Title: Chronic Effect of Cardiorespiratory Training on Ventilatory Muscle Strength in Elderly Women: Controlled Trial, Randomized and Double Blind.
Brief Title: Cardiorespiratory Training and Ventilatory Muscle Strength
Acronym: RMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Gama Filho (Other)
Responsible Party: Principal Investigator, Fabio Dutra Pereira, Chronic effect of cardiorespiratory training on ventilatory muscle strength in elderly women: Experiment controlled, randomized and double blind., Universidade Gama Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR20132014
Record Dates: First submitted 2013-06-03; First posted 2013-07-31 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cardiorespiratory training (Experimental): The cardiorespiratory training group will undergo 18 sessions, these also periodized in a maximum six weeks, respecting the minimum weekly frequency of 3 sessions.
  Interventions: Other: Cardiorespiratory training
- Ventilatory Training (Active Comparator): The ventilatory training group will undergo 18 sessions, periodized in a maximum six weeks, respecting the minimum weekly frequency of three sessions.
  Interventions: Other: ventilatory training
- Crontrol Group (No Intervention): This condition will last six weeks, this period will be held six lectures sixty minutes long and periodization weekly.

INTERVENTIONS:
Other: Cardiorespiratory training — The cardiorespiratory training group will undergo 18 sessions, these also periodized in a maximum six weeks, respecting the minimum weekly frequency of 3 sessions.
  Other Names: GTC
  Arms: Cardiorespiratory training
Other: ventilatory training — The ventilatory training group will undergo 18 sessions, periodized in a maximum six weeks, respecting the minimum weekly frequency of three sessions.
  Other Names: GTV
  Arms: Ventilatory Training

SUMMARY:
The cardiorespiratory training can increase muscle strength ventilatory.

DETAILED DESCRIPTION:
Specifically for being an experiment parallel factorial intervention after met the eligibility criteria for the participants will be randomly allocated to three groups: control, respiratory training, cardiorespiratory training (indoor Bike).

ELIGIBILITY:
Inclusion Criteria:

- Have lower maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) values normative reference proposed by the Brazilian Society of Thoracic.

Exclusion Criteria:

* Not be voluntary to the present study.
* Conditions that oblige participants are absent for more than two weeks of activities performed in the experiment.

Ages: 60 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Ventilatory muscle strength | The ventilatory muscle strength (MIP and MEP) will be measured after 18 cardiorespiratory training sessions held in 6 weeks.
  The MIP and MEP are measured by a digital manometer 300(BRAZIL). During the measurement the participants should be seated in a chair type office allowing your upper body to remain in contact with the back of it, forming an angle of 90° to the hip, the arms extended along the body, knees flexed too 90° and feet flat on the floor. Participants will use a nose clip.
  The evaluator will manually compress the face of the participant not allowing the contraction of the buccinator muscles increase intraoral pressure and interfere with the measurement result.
  In the measurement of MIP participants should hold a maximum inspiration from residual volume (RV) and MEP maximum exhalation from total lung capacity (TLC).

CONTACTS AND LOCATIONS:
Overall Officials: Fabio D Pereira, MSc, Principal Investigator — Gama Filho University
Locations (1):
- Gama Filho University, Rio de Janeiro, Rio de Janeiro, Brazil